CLINICAL TRIAL: NCT04983667
Title: Supplementation of Zinc-AA Complexes in Women During Pregnancy and Lactation, to Assess Effects on Autism Spectrum Disorder (ASD), Immune Status and Gut Microbiota in Offspring
Brief Title: Zinc-AA Supplementation During Pregnancy & Lactation to Assess Effects on ASD Prevalence in Offspring
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: A funding agreement could not be secured with the primary funding organizations
Sponsor: Instituto Tecnologico y de Estudios Superiores de Monterey (Other)
Responsible Party: Principal Investigator, Victor Javier Lara-Diaz, M.D., Ph.D., Professor-Researcher, Instituto Tecnologico y de Estudios Superiores de Monterey
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Zinc-Autismo
Record Dates: First submitted 2021-07-11; First posted 2021-07-30 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Autism Spectrum Disorder; Zinc Deficiency; Pregnancy Related
Keywords: Zinc supplementation; Pregnancy
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Parallel 1:1 randomization to one of two interventions, the active compound or the placebo
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Randomized allocation to one of two supplements, one has the active compound, the other is a placebo. Identical containers and labels have been designed. Both groups will receive the customary iron sulfate and folic acid supplementation along pregnancy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orange (Experimental): Zinc-AA, Tablet, 30 mg. PO, Once Daily for up to one year
  Interventions: Dietary Supplement: Zn-AA
- Green (Placebo Comparator): Placebo, Tablet, 30 mg. PO, Once Daily for up to one year.
  Interventions: Dietary Supplement: Zn-AA

INTERVENTIONS:
Dietary Supplement: Zn-AA — Oral supplementation of either 30 mg daily or Zinc-AA complex or placebo, from the study recruitment during first trimester of pregnancy, all through pregnancy and up to the sixth month after giving birth.

SUMMARY:
Autism and associated entities, grouped under the Autism Spectrum Disorders (ASD) is the fastest growing intellectual disability in the world, statistics signal for a 1 to 3% prevalence on infants. The cause is unknown, although some data suggest that zinc deficiency during pregnancy may have an important role in its presentation. This study seeks to supplement the nutrition of randomly selected prospective and actually pregnant women with a zinc-Amino-acid complex (Zn-AA), during pregnancy and early lactation, and compare the rate of ASD in their offspring with the rate in a similar and also randomly selected cohort of non supplemented women, to assess if Zn-AA supplementation during pregnancy has any effect on this outcome

DETAILED DESCRIPTION:
Autism and associated disorders (Autism Spectrum Disorders, ASD) is the fastest growing disability in the world, statistics indicate a prevalence of between 1 and 3%. This entity is the one that generates more stress in families, four times more than in a neuro-typical family and twice more than in a family with any other disability. Besides, this condition increases health spending for the family, the state and the country.

By not knowing the cause, and witnessing the growth of this disability, with the prevalence described, and the births reported in 2019 in Mexico (2,092,214), we expect between 20,922 and 62,766 new cases in our country each year. In Nuevo León, a state in the northeast of Mexico, the average birth rate per year from 2017 to 2019 (latest official data available) is 91,484, which makes us estimate an incidence of 915 to 2744, for the same period. ASD is also a family stressful disability, associated to a high rate of separations, social isolation and divorces, which leads to social problems of alarming dimensions. In the United States, for 2025 the cost of Autism is projected at 1 trillion dollars, associated with medications, interventions and educational expenses.

In Mexico, the lack of universal diagnostic screening, detection and intervention programs before the age of three years makes those affected to require important support throughout their lives, since the benefits of early intervention are lost.

This project consists of two parts. The first is the Primary Study. It consists of establishing whether the supplementation of Zinc-AA complexes, in women during pregnancy and lactation, has any effect on the prevalence of Autism and if it favorably modifies the immunological and metabolic status of the mother and the progeny; seeks to confirm the findings that our group of investigators has obtained in published pre-clinical investigations that found that a Zinc deficiency in the mother (mice and human erythrocytes), caused by dietary factors, provokes changes in the morphology of the intestine of the progeny, as well as modifications in the microbiota and increased inflammatory markers in the blood and brain, similar to those reported in people with Autism. In Latin America, the diet is based on cereals, and i so abundant in dietary fiber and phytates. These factors, along supplements usually recommended to mothers who plan to become pregnant (Calcium, Iron and Folic Acid), predispose these women to Zinc deficiency. We are also proposing a Secondary Study, to establish the zinc status and the characteristics of the intestinal microbiome in young, non-pregnant adult women, as a comparative reference standard.

Until now, there are no projects in the world that seek to partially or totally solve the causes of Autism, this is the first study that seeks to prevent the problems associated with autism and could be the first to influence the reduction of the incidence of Autism. This project will involve Mexican researchers from Instituto Tecnologico y de Estudios Superiores de Monterrey (ITESM), as well as researchers from the University of Limerick, Ireland, from the University Clinic of the Autonomous University of Nuevo León, in the northeast of Mexico; as well as the Laboratory of Dr. Fanis Missirlis, of the National Polytechnic Institute, in Mexico City.

This project has the financial support of the International Zinc Association (IZA), managed by Zinpro Corp., represented in Mexico by Elemend Salud, representative Ing. Guillermo Vela Staines (g.vela@zinpro.com).

ELIGIBILITY:
Inclusion Criteria:

* Women from 18 to 35 years of age, pregnant, within the 12th and 20th week (Primary study) or with the intention to get pregnant in the following six months (Secondary study)
* Hemoglobin over 8 g/dL
* Accepting to be included in a standard pediatric physical and neurobehavioral follow-up program from birth and to at least 18 months of age.
* Accepting to receive the Zinc supplement (or placebo) and to ingest it daily from the inclusion to the study and up to the sixth postnatal month
* Agreement to read and sign the Informed Consent Document

Exclusion Criteria:

* Women who do not accept to deliver in a hospital setting, or without immediate access to a proper facility
* Women with self-reported alcohol or drug addiction
* Women with a sero positivity to HIV, even if under treatment
* Women with a pregnancy resulted from assisted or in vitro fertilization techniques
* Women with an active severe acute respiratory syndrome-Coronavirus (SARS-CoV2) infection

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-23 (Actual)

PRIMARY OUTCOMES:
Autism spectrum disorder | From 16 to 20 months of age
  Positive identification of any component of the Autism Spectrum Disorder (ASD) through the Autism Diagnosis Observation Schedule, 2nd edition (ADOS-2) specialized battery of tests, which provide a standardized set of tests that offer as output a set of ranges of concern reflecting the extent to which a child demonstrates behaviors associated with ASD.

SECONDARY OUTCOMES:
Microbiota modification associated to maternal zinc supplementation or placebo during pregnancy | From birth to six months of age
  Comparative analysis of the microbiome composition (Type and relative quantity of micro-organisms) in a subset of the supplemented and the un-supplemented groups, at birth, and also at the end of the first six months of lactation
Immune phenotype | From birth to six months of age
  Comparison of the Immune phenotype (Type and quantity of main Interleukines and Cytokines in peripheral blood, and characterization of Leucocyte population and subpopulation, also in peripheral blood) in a subset of the supplemented and the un-supplemented groups, at birth, and also at the end of the first six months of lactation

CONTACTS AND LOCATIONS:
Overall Officials: Rebeca Thelma Martínez-Villarreal, M.D., Ph:D., Principal Investigator — Universidad Autónoma de Nuevo León, Centro Universitario de Salud, Campus de la Salud
Locations (1):
- Centro Universitario en Salud, San Nicolás de los Garza, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Data will be archived in the Institutional Repository
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: One year upon completion
Access Criteria: To qualified health researchers upon request, all data will be anonymized.